CLINICAL TRIAL: NCT04894929
Title: Comprehensive Geriatric Assessment in the Monitoring of Functional Improvement Through Vestibular and Multicomponent Exercises.
Brief Title: Comprehensive Geriatric Assessment in the Monitoring of Functional Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, MARINA LOPEZ GARCIA, Associated Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Useville2
Record Dates: First submitted 2021-05-09; First posted 2021-05-20 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Aging; Vestibular Disorder; Physiotherapy; Physical Activity
Keywords: aging, physiotherapy, physical activity, balance
MeSH Terms: conditions — Vestibular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: set of interventions can be carried out by making an initial diagnosis of pre-frailty or frailty using instruments and simple validated tests. This is indicated or thus recommended in the guidelines from national and international societies (24-25). In this sense, we can use a comprehensive assessment of the VALINTAN (computerized) tool, a VGI-type assessment, whose axis is function, focusing on predefined diagnoses associated with effective documented interventions or with functional fragility or loss. Currently the tool is open and freely accessible (26).
Who Masked: Participant
Masking Description: It has been explained to the patient that the exercises that they are going to perform are going to serve for their functional improvement, but the exercises are different depending on the group to which they have been assigned randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A. Multi-conponente exercise (Experimental): 1. A 6-week therapeutic multi-component physical exercise program will be carried out. The ministerial guide will be followed by carrying out 5 weekly sessions (from Monday to Friday), offering the application through a web link of the weekly programming of the exercises for the patient (type of exercise, video of its execution, number of repetitions and description) having a approximate duration of 40 minutes.
  2. Said sessions will be carried out daily and from the center a call was made at the end of the week to mark the follow-up and resolve any questions related to symptoms
  Interventions: Other: multi component exercise in the clinic; Other: multi component exercise at home telerehabilitation
- B. Vestibular exercise (Experimental): The vestibular exercises will be performed with the instructions of a physiotherapist, in sessions of about 20 minutes with 5 weekly sessions (Monday to Friday) consisting of 5 repetitions without fatigue of:
  to. Head and eye movements while sitting. b. Head and body movements while sitting. c. Exercises standing. d. Combined exercises of modifications in steps, unstable surfaces and in progress.
  and. Along with push up 30sec and squat 30sec All participants will have a weekly follow-up from Monday to Friday to control attendance and compliance via telephone.
  Interventions: Other: vestibular exercise in the clinic; Other: vestibular exercise at home telerehabilitation

INTERVENTIONS:
Other: multi component exercise in the clinic — Patients randomly assigned to this group have a pre-fragile or fragile SPPB condition, so they will perform:
  3 days of empowerment work, 4 days of flexibility work, and daily walking aerobic work and balance work.
  Arms: A. Multi-conponente exercise
Other: vestibular exercise in the clinic — Patients randomly assigned to this group have a pre-fragile or fragile SPPB condition, so they will perform. sessions of about 20 minutes with 5 weekly sessions (Monday to Friday) consisting of 5 repetitions without fatigue of:
  to. Head and eye movements while sitting. b. Head and body movements while sitting. c. Exercises standing. d. Combined exercises of modifications in steps, unstable surfaces and in progress.
  and. Along with push up 30sec and squat 30sec
  Arms: B. Vestibular exercise
Other: vestibular exercise at home telerehabilitation — Patients randomly assigned to this group have a pre-fragile or fragile SPPB condition, so they will perform with the help of a video. sessions of about 20 minutes with 5 weekly sessions (Monday to Friday) consisting of 5 repetitions without fatigue of:
  to. Head and eye movements while sitting. b. Head and body movements while sitting. c. Exercises standing. d. Combined exercises of modifications in steps, unstable surfaces and in progress.
  and. Along with push up 30sec and squat 30sec
  Arms: B. Vestibular exercise
Other: multi component exercise at home telerehabilitation — Patients randomly assigned to this group have a pre-fragile or fragile SPPB condition, so they will perform with the help of a video:
  3 days of empowerment work, 4 days of flexibility work, and daily walking aerobic work and balance work.
  Arms: A. Multi-conponente exercise

SUMMARY:
14.44% of the Spanish population is over 70 years old and Aging as a normal process is characterized by gradual modifications in the physiological functions of the different systems, so that as age progresses, deterioration can lead to imbalances and alterations in health that cause diseases or traumatic processes. Within these processes, vestibular loss occurs normally in the face of healthy aging and, encompassed within this progressive dysfunction, various symptoms such as dizziness, imbalances, facial and limb weakness, confusion or headache may occur.

Functional status is the best indicator of the overall health status of the elderly person. Identifying these indicators as soon as possible is the best way to prevent functional decline and promote active aging and life expectancy free of disability. For this reason, there are strategies that are currently a priority in health systems. The special COVID circumstances eliminate the possibility of group work and invite the realization at home or individually of workshops or collective exercises In the field of physiotherapy, vestibular exercises have shown efficacy for improving balance and reducing the risk of falls in cognitively intact people without vestibular impairment, being a specific approach to vestibular rehabilitation for the reduction of dizziness and imbalances , as it facilitates the compensation of the Central Nervous System. physiotherapy intervention has been shown in various studies to be effective in improving balance and reducing the risk of falls in older people.

Also considering that the control of body balance in the elderly depends not only on the vestibular system, but also on the correlations between all the other systems, it seems interesting to add exercises with multiple components, since it would add effects of improvement in functional independence of people greater for daily activities and control of body balance.

Therapeutic physical exercise is an effective non-pharmacological strategy to improve the functional condition of the elderly and although it is known that there are various exercise modalities that improve physical function and quality of life, The Clinical Practice Guidelines emphasize the importance of multicomponent / multimodal exercise for this population group

DETAILED DESCRIPTION:
Therefore, and given the information in both directions, we consider that it is necessary to determine the efficacy in the evidence of both actions (multicomponent exercise and vestibular exercises) to improve functional capacity and thus prevent falls, conducting a randomized clinical trial that compares the effectiveness of both interventions. Given the special circumstances during the COVID-19 pandemic, an online or virtual follow-up is necessary to achieve the exercises, building a resource website and helping virtual access and monitoring to carry out the personalized exercise.

Thus, this set of interventions can be carried out by making an initial diagnosis of pre-frailty or frailty using instruments and simple validated tests. This is indicated or recommended in the guidelines from national and international societies. In this sense, we can avail ourselves of a comprehensive assessment of the VALINTAN tool (computerized comprehensive assessment of the elderly and used in primary care), whose axis is function, focuses on predefined diagnoses associated with effective documented interventions or with the fragility or functional loss. Currently the tool is open and freely accessible

ELIGIBILITY:
Inclusion Criteria:

1. Women and men over 70 years old.
2. Having assessed through the VALINTAN (online free tool in primary care por comprehensive assessment of the elderly) of function their integral functional status and determining as a health process deterioration functional and lack of physical activity.
3. Subjects with a score between 4 and 9 points according to the "Short Physical Performance Battery" (SPPB) scale

Exclusion Criteria:

- 1) patients without gait independence or who did not pass the previous evaluation in SPPB.

2) Polypharmacological patients (combined use of beta-blockers, sulpiride or betahistine) will also be considered for exclusion.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Barthel test | _measure 1: before start treatment _Measure 2: up to 6 weeks (after treatment)
  balance
VIDA test | _measure 1: before start treatment _Measure 2: up to 6 weeks (after treatment)
  Questionnaire for Instrumental Activities of Daily Living (AIVD)
short Performance Physical Battery (SPPB) | _measure 1: before start treatment _Measure 2: up to 6 weeks (after treatment)
  Gait capacity: SPPB physical function assessment battery

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Suárez Serrano, PT, Study Director — University of Seville
Locations (1):
- Fundomar Elderly nursing home, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
The intention is to publish in an impact magazine

REFERENCES:
- [Background] Kularbpthettong K. Effects of the Physical Therapy Application for Elderly. Advances in Intelligent Systems and Computing. 2020 Vol 1152: 462-467
- [Result] Iwasaki S, Yamasoba T. Dizziness and Imbalance in the Elderly: Age-related Decline in the Vestibular System. Aging Dis. 2014 Feb 9;6(1):38-47. doi: 10.14336/AD.2014.0128. eCollection 2015 Feb. PMID 25657851
- [Result] Agrawal Y, Carey JP, Della Santina CC, Schubert MC, Minor LB. Disorders of balance and vestibular function in US adults: data from the National Health and Nutrition Examination Survey, 2001-2004. Arch Intern Med. 2009 May 25;169(10):938-44. doi: 10.1001/archinternmed.2009.66. PMID 19468085
- [Result] Agrawal Y, Zuniga MG, Davalos-Bichara M, Schubert MC, Walston JD, Hughes J, Carey JP. Decline in semicircular canal and otolith function with age. Otol Neurotol. 2012 Jul;33(5):832-9. doi: 10.1097/MAO.0b013e3182545061. PMID 22699991
- [Result] Brown KE, Whitney SL, Marchetti GF, Wrisley DM, Furman JM. Physical therapy for central vestibular dysfunction. Arch Phys Med Rehabil. 2006 Jan;87(1):76-81. doi: 10.1016/j.apmr.2005.08.003. PMID 16401442
- [Result] Klatt BN, Ries JD, Dunlap PM, Whitney SL, Agrawal Y. Vestibular Physical Therapy in Individuals With Cognitive Impairment: A Theoretical Framework. J Neurol Phys Ther. 2019 Apr;43 Suppl 2(Suppl 2 Spec INTERNATIONAL CONFERENCE ON VESTIBULAR REHABILITATION):S14-S19. doi: 10.1097/NPT.0000000000000266. PMID 30883488
- [Result] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496
- [Result] Howe TE, Rochester L, Neil F, Skelton DA, Ballinger C. Exercise for improving balance in older people. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD004963. doi: 10.1002/14651858.CD004963.pub3. PMID 22071817
- [Result] Swanenburg J, Wild K, Straumann D, de Bruin ED. Exergaming in a Moving Virtual World to Train Vestibular Functions and Gait; a Proof-of-Concept-Study With Older Adults. Front Physiol. 2018 Jul 31;9:988. doi: 10.3389/fphys.2018.00988. eCollection 2018. PMID 30108511
- [Result] Martins E Silva DC, Bastos VH, de Oliveira Sanchez M, Nunes MK, Orsini M, Ribeiro P, Velasques B, Teixeira SS. Effects of vestibular rehabilitation in the elderly: a systematic review. Aging Clin Exp Res. 2016 Aug;28(4):599-606. doi: 10.1007/s40520-015-0479-0. Epub 2015 Oct 28. PMID 26511625
- [Result] Macias JD, Massingale S, Gerkin RD. Efficacy of vestibular rehabilitation therapy in reducing falls. Otolaryngol Head Neck Surg. 2005 Sep;133(3):323-5. doi: 10.1016/j.otohns.2005.04.024. PMID 16143174
- [Result] Beato M, Dawson N, Svien L, Wharton T. Examining the Effects of an Otago-Based Home Exercise Program on Falls and Fall Risks in an Assisted Living Facility. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):224-229. doi: 10.1519/JPT.0000000000000190. PMID 29698252
- [Result] Fishleder S, Petrescu-Prahova M, Harris JR, Leroux B, Bennett K, Helfrich CD, Kohn M, Hannon P. Predictors of Improvement in Physical Function in Older Adults in an Evidence-Based Physical Activity Program (EnhanceFitness). J Geriatr Phys Ther. 2019 Oct/Dec;42(4):230-242. doi: 10.1519/JPT.0000000000000202. PMID 29979352
- [Result] Bean JF, Brown L, DeAngelis TR, Ellis T, Kumar VSS, Latham NK, Lawler D, Ni M, Perloff J. The Rehabilitation Enhancing Aging Through Connected Health Prehabilitation Trial. Arch Phys Med Rehabil. 2019 Nov;100(11):1999-2005. doi: 10.1016/j.apmr.2019.04.015. Epub 2019 May 29. PMID 31152705
- [Result] Canli S, Ozyurda F. A multi-modal exercise intervention that improves cognitive function and physical performance, elderly with mobility-related disability: a randomized controlled trial. J Sports Med Phys Fitness. 2020 Jul;60(7):1027-1033. doi: 10.23736/S0022-4707.20.10286-X. Epub 2020 Apr 6. PMID 32253894
- [Result] Martin Lesende I, Mendibil Crespo LI, Berrizbeitia Gonzalez A, Llamosas Luengo I. [Computerized geriatric assessment tool VALINTAN (www.valintan.com) for primary care]. Aten Primaria. 2020 Oct;52(8):590-591. doi: 10.1016/j.aprim.2020.04.016. Epub 2020 Jun 15. No abstract available. Spanish. PMID 32553538
- [Result] de Hoyos Alonso MDC, Gorronogoitia Iturbe A, Martin Lesende I, Baena Diez JM, Lopez-Torres Hidalgo J, Magan Tapia P, Acosta Benito MA, Herreros Herreros Y; Grupo de Actividades Preventivas en los Mayores del PAPPS. Actividades preventivas en los mayores. Actualizacion PAPPS 2018. Aten Primaria. 2018 May;50 Suppl 1(Suppl 1):109-124. doi: 10.1016/S0212-6567(18)30365-2. No abstract available. Spanish. PMID 29866352
- See also: Consensus document on prevention of frailty and falls in the elderly. SPAIN. Health Promotion and Prevention Strategy in the SNS Document approved by the Inter-territorial Council of the National Health System on June 11, 2014. Ministry of Health, Social — https://www.sanidad.gob.es/areas/promocionPrevencion/envejecimientoSaludable/fragilidadCaidas/estrategiaSNS/home.htm
- See also: SPAIN. National Institute of Statistics [Internet database]. — https://www.ine.es/